CLINICAL TRIAL: NCT00024479
Title: Studies of the Natural History of Rheumatic Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010227; 01-AR-0227
Record Dates: First submitted 2001-09-14; First posted 2001-09-14 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Rheumatic Diseases; Arthritis
Keywords: Minorities; Rheumatic Disease; Community Based; Natural History; Ethnicity; Health Disparities
MeSH Terms: conditions — Rheumatic Diseases; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspected or confirmed rheumatic disease: autoimmune, autoinflammatory, or degenerative conditions

SUMMARY:
This study will explore the causes of rheumatic diseases and why many of them affect certain minority communities more severely. Rheumatic diseases may cause joint pain, stiffness or swelling. Some can involve bones, muscles, tendons or ligaments. Some cause abnormalities of the immune system-the body s defense against disease. Some rheumatic diseases are painful or deforming and some can be life threatening. Information obtained from this study will be used to learn about the disparities in rheumatic disease in the minority community and to design further, more targeted, research studies to address this issue.

Patients with known or suspected rheumatic disease 18 years of age or older may be eligible for this study. Candidates will undergo a medical history and physical examination to confirm the diagnosis of rheumatic disease and determine what is needed for evaluation and treatment.

Participants will receive standard medical care for rheumatic disease and arthritis. No experimental treatments, medications or procedures will be included in this study. Procedures may include routine blood tests for blood chemistries, cell counts, and antibodies commonly found in patients with rheumatic disease; a urine test for proteins and cells; and X-rays and other imaging tests to check for abnormalities in the lungs or other organs. All medical information will be kept confidential.

Patients who are found to be eligible for other current NIH research studies will be offered an opportunity to participate in these studies.

DETAILED DESCRIPTION:
This protocol will permit the evaluation and treatment of subjects who are members of the minority community, for the purpose to facilitate understanding the pathogenesis and natural history of rheumatic diseases in this community. Patients will be evaluated with a history and physical examination and routine laboratory studies will be obtained as needed to assess diagnosis, disease activity, disease complications and to monitor for treatment-related responses and toxicities. Patients eligible for other research protocols will be offered an opportunity to participate in these studies by signed informed consent. Any medical care recommended or provided to the patient will be consistent with routine standards of practice and will be provided in consultation with the patient s referring physician. All patients referred to this study must have a health care provider provide a referral. The establishment of this protocol will provide a means to evaluate and treat patients from the minority community, and to generate hypotheses and protocols based on this clinical experience that will address questions of health disparities in the rheumatic diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Known or suspected rheumatic disease

Age greater than or equal to 18 years

Willingness and capacity to provide informed consent.

EXCLUSION CRITERIA:

Patients will be excluded if any of the inclusion criteria cannot be met.

Women who are pregnant or breastfeeding at the time of enrollment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, older than or equal to 18 years of age, referred from the community
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2001-10-03 (Actual)

PRIMARY OUTCOMES:
To generate hypotheses relating to the basis and/or effects of health disparities in the community, which may serve as the basis for subsequent research efforts based in the community and/or at the NIH Clinical Center | 31 Years
  The rheumatological health of the community

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The protocol is silent on IPD.

REFERENCES:
- [Background] Reveille JD, Moulds JM, Ahn C, Friedman AW, Baethge B, Roseman J, Straaton KV, Alarcon GS. Systemic lupus erythematosus in three ethnic groups: I. The effects of HLA class II, C4, and CR1 alleles, socioeconomic factors, and ethnicity at disease onset. LUMINA Study Group. Lupus in minority populations, nature versus nurture. Arthritis Rheum. 1998 Jul;41(7):1161-72. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-K. PMID 9663471
- [Background] Lawrence RC, Helmick CG, Arnett FC, Deyo RA, Felson DT, Giannini EH, Heyse SP, Hirsch R, Hochberg MC, Hunder GG, Liang MH, Pillemer SR, Steen VD, Wolfe F. Estimates of the prevalence of arthritis and selected musculoskeletal disorders in the United States. Arthritis Rheum. 1998 May;41(5):778-99. doi: 10.1002/1529-0131(199805)41:53.0.CO;2-V. PMID 9588729
- [Background] Jordan JM. Effect of race and ethnicity on outcomes in arthritis and rheumatic conditions. Curr Opin Rheumatol. 1999 Mar;11(2):98-103. doi: 10.1097/00002281-199903000-00003. PMID 10319211
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-AR-0227.html